CLINICAL TRIAL: NCT02686736
Title: Evaluation of the Effect of an Internet-based Educational Intervention to Prevent Risky Sexual Behaviors in Mexican Adolescents
Brief Title: Internet-based Intervention to Prevent Risky Sexual Behaviors in Mexican Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: Hospital Infantil de Mexico Federico Gomez (Other); Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Principal Investigator, Svetlana Doubova, Head of the Epidemiology and Health Services Research Unit, Coordinación de Investigación en Salud, Mexico
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R 2014-785-033
Record Dates: First submitted 2016-02-11; First posted 2016-02-19 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Adolescent Behavior
Keywords: internet-based educational intervention; risky sexual behaviors; prevention
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet-based educational intervention (Other): The Internet-based educational intervention will include four educational sessions that will be provided during a four-week period. The follow up will last three-months.
  Interventions: Behavioral: Internet-based educational intervention
- Control group (No Intervention): In the control group, teens will continue the usual school provided sexual education and will be invited to answer the internet-based self-applied questionnaire at the same time as the intervention group.

INTERVENTIONS:
Behavioral: Internet-based educational intervention — The intervention will include four educational sessions about risky sexual behaviors and its prevention. The intervention will last one month (one session per week) followed by a three-month follow-up. Teens will be allowed to access to a weekly session at any time and as often as he/she likes.
  Arms: Internet-based educational intervention

SUMMARY:
The objective of this study is to design and evaluate an internet-based educational strategy to prevent sexual risk behaviors in Mexican adolescents. Methods: A field trial with one intervention and one comparison group, with ex-ante and ex-post measurements will be conducted in 2 public secondary schools. Adolescents between 14 and 15 years of age will participate. The intervention will be conducted in one school and the other school will serve as a comparison group, where investigators will observe the usual sexual education that the school provides. The intervention will be delivered through an internet web page; it includes four educational sessions that will be provided during a four-week period. The follow up will last three-months. The information on the study variables will be obtained through an internet-based self-applied questionnaire and collected on three occasions: when the adolescents enters to the study (baseline), once intervention is completed (at one month) and after three months of follow-up (at fourth month).

DETAILED DESCRIPTION:
The conceptual framework for the intervention and educational materials was based on the model of the Information-Motivation-and-Behavioral-Skills proposed by Fisher and Fisher, 2000. This model emphasizes that adequate information regarding risk sexual behavior, changing the motivational component and training in behavioral skills can influence initiation and maintenance of protective sexual behaviors.

The research group that was constituted by a pediatrician, a psychologist, and a sociologist, designed the educational materials. All the research team members have experience in educational interventions. The academic basis to develop the materials were two books titled: "You, your life, your dreams" developed by International Family Care (2007) and "Your future in freedom, for responsible sexuality and reproductive health" published by the Government of the Federal District and the Secretary of Education of the Federal District of Mexico City (2008). Investigators also took into account the statistics on the sexually transmitted diseases and adolescents' pregnancies of the World Health Organization, 2012 National Health and Nutrition survey, the National Register of AIDS cases, and information from the Planned Parenthood Federation of America.

Investigators designed teen-friendly educational materials, to do so, investigators used "avatars" from www.bitstrips.com, which are the comics for teenagers. Investigators created two central characters a teenage boy and a teenage girl who present the information in the form of dialogs and talk about their own and friend's experiences.

Two experts in the area of adolescents' sexual and reproductive health reviewed the educational materials; then, 20 adolescents between 14 and 15 years participated in three rounds of pilot testing. Both, the teenagers and their parents accepted to participate in this phase through verbal informed consent.

Investigators used the snowball sampling technique to choose the teenagers that took part in the pilot phase, which included ten boys and ten girls, with an average grade point of 8.5 (range 8.0-9.0). Their families were of different types (nuclear, single-parent, extended), and their parents had varying levels of education. Most adolescents (18) had not begun sexual activity, and only two reported being sexually active. Experts and teens were asked if the educational information was clear, understandable and if it used appropriate language for teens, or if it was contradictory, uncomfortable, or boredom. The teens were asked to evaluate whether they liked or not each educational session (using a scale of 1 to 3, where 1 = No, I do not like it, 2 = I like it more or less, 3 = I like it) and to explain why they disliked the educational information. The final version of the educational material was produced taking into account the comments and suggestions of experts and teens, which rated the information highly. Although most adolescents who participated in the pilot testing had not started their sexual life, they reported that the information was clear and interesting.

Description and evaluation of the intervention The study materials are available on the Internet web page (http://tu-ssexual.com), which can be accessed with the participant e-mail address and a centrally assigned password.

The intervention will include an introduction and four educational sessions and will last one month (one session per week) followed by a three-month follow-up. Teens will be allowed to access to a weekly session at any time and as often as he/she likes. However, the sessions will be consecutive, so teens cannot be able to access to the next session without finishing the previous one. Each session has the duration of one hour on average and ends with overview questions. Additionally, at the end of the each session teens will be asked ¿what they like and dislike about the session? And the answers will be recorded in the study database.

Furthermore, during the intervention and follow-up booster e-mail messages will be sent to the teens of the intervention group. "Booster messages" will emphasize main points of the educational sections and will be sending 2-3 per week from the second week of the intervention.

Information on the study variables will be obtained through the internet-based self-applied questionnaire and collected on three occasions: when the adolescents enters into the study (baseline), once the intervention is completed (at one month) and after three months of follow-up (fourth month).

ELIGIBILITY:
Inclusion Criteria:

* Adolescents between 14 and 15 years of age, who are in the third year of public secondary schools and attend to schools that were selected through simple random sampling from the list of public secondary schools in the Iztapalapa Delegation in Mexico City
* Who agree to participate through informed consent; also, their parents must sign the written informed consent.

Exclusion Criteria:

* None

Ages: 14 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 456 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in attitudes regarding condom use at 1 and 4 months measured by the University of California, Los Angeles Multidimensional Condom Attitudes Scale | Baseline, 1 month, and 4 months
  Attitudes regarding condom use will be measured by the University of California, Los Angeles Multidimensional Condom Attitudes Scale.

SECONDARY OUTCOMES:
Change from baseline in knowledge of sexually transmitted infections at 1 and 4 months measured by the scale validated in Mexican teens by Robles-Montijo and Diaz-Loving | Baseline, 1 month, and 4 months
  Knowledge of sexually transmitted infections will be measured by the scale validated in Mexican teens by Robles-Montijo and Diaz-Loving.
Change from baseline in self-efficacy toward consistent condom use at 1 and 4 months assessed by the seven measures proposed by Fishbein and colleagues | Baseline, 1 month, and 4 months
  Self-efficacy toward consistent condom use will be assessed by the seven measures proposed by Fishbein and colleagues.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Doubova SV, Martinez-Vega IP, Infante-Castaneda C, Perez-Cuevas R. Effects of an internet-based educational intervention to prevent high-risk sexual behavior in Mexican adolescents. Health Educ Res. 2017 Dec 1;32(6):487-498. doi: 10.1093/her/cyx074. PMID 29177452
- [Derived] Doubova SV, Infante-Castaneda C, Perez-Cuevas R. Internet-based educational intervention to prevent risky sexual behaviors in Mexican adolescents: study protocol. BMC Public Health. 2016 Apr 18;16:343. doi: 10.1186/s12889-016-2990-4. PMID 27089870